CLINICAL TRIAL: NCT03119519
Title: Local Non-salvage Radiotherapy for Synchronous Oligometastatic Non-small-cell Lung Cancer :A Multicenter,Randomized,Controlled,Phase 2 Study.
Brief Title: Local Non-salvage Radiotherapy for Synchronous Oligometastatic Non-small-cell Lung Cancer.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Southern Medical University, China (Other)
Responsible Party: Principal Investigator, Xiaoxia Zhu, Professor, Southern Medical University, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LC2019ZD009
Record Dates: First submitted 2017-04-13; First posted 2017-04-18 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Stage IV Non-small Cell Lung Cancer
Keywords: NSCLC; Oligometastases; radiotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Intervention Model Description: A randomized phase II trial of first line chemotherapy or targeted therapy plus local definitive radiotherapy or not for patients with synchronous oligometastatic non-small cell lung cancer
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Local Definitive Radiotherapy (Experimental): Standard platinum-based doublet chemotherapy or EGFR-TKI (Gefitinib or Erlotinib) followed by 3D-CRT (three-dimensional conformal radiotherapy) or IMRT (intensity modulated radiotherapy) to primary thoracic foci or remediable oligometastatic focus.
  Interventions: Radiation: Local Definitive Radiotherapy; Drug: No Local Definitive Radiotherapy
- No Local Definitive Radiotherapy (Active Comparator): Standard platinum-based doublet chemotherapy or EGFR-TKI (Gefitinib or Erlotinib) alone, according to gene test.
  Interventions: Drug: No Local Definitive Radiotherapy

INTERVENTIONS:
Radiation: Local Definitive Radiotherapy — three-dimensional conformal therapy or intensity modulated radiation therapy
  Other Names: LDR
  Arms: Local Definitive Radiotherapy
Drug: No Local Definitive Radiotherapy — Standard platinum-based doublet chemotherapy or EGFR-TKI (Gefitinib or Erlotinib) alone, according to gene test.
  Other Names: Non-LDR

SUMMARY:
Aggressive therapy may improve survival in synchronous oligometastatic NSCLC and the goal of this clinical trial is to assess the efficacy and safety of local definitive radiotherapy in this subset of patients.

DETAILED DESCRIPTION:
For NSCLC patients with synchronous oligometastases, first line chemotherapy or targeted therapy concurrent with non-salvage radiotherapy on metastatic or primary thoracic tumor contributed a longer progression-free survival than chemotherapy or targeted therapy alone.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 18 to 70 years old;
2. Histologically or cytologically confirmed non-small cell lung cancer;
3. Stage IV patients with measurable primary tumor and distant metastases number ≤5；
4. PS score 0-2；
5. Have never received local or systemic anti-cancer treatment, including surgery (biopsy is allowed), first line chemotherapy, targeted therapy or immunotherapy;
6. Life expectancy of >3 months;
7. Organ function levels must meet the following requirements:

(1)Bone marrow: White blood cell (WBC)≥4.0G/L；neutrophile granulocyte (NEU)≥1.5G/L；platelets (PLT)≥100G/L; hemoglobin (HGB)≥9g/L； (2)Liver and kidney: total bilirubin (TBIL), aspartate aminotransferase (AST), alanine aminotransferase (ALT)≤2.0 × the upper limit of normal (ULN)；creatinine≤1.5×ULN; 8.Patient must be willing and able to provide written informed consent.

Exclusion Criteria:

1. The amount of metastatic focus >5;
2. Patient can't tolerate chemotherapy or targeted therapy;
3. Local or systemic anti-cancer treatment had been used for the primary foci and metastatic lymph nodes, including surgery (biopsy is allowed), first line chemotherapy, targeted therapy or immunotherapy;
4. Previous or concurrent suffered from other malignancies;
5. Concurrent with other serious disease that can not be controlled;
6. Women who are breast-feeding or pregnant;
7. Have an allergy to pemetrexed, cisplatin, taxanes, targeted medicine and contrast agent;
8. Patients with poor obedience or researchers think that the patient may not be able to accomplish the whole trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2017-12-11 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) | 5 years
  Refers to the time from randomization to disease progression or death.

SECONDARY OUTCOMES:
Local tumor control | up to 5 years
  From time of randomization to time of progression or death（according to RECIST v1.1 [）
Oligometastatic foci control | up to 5 years
  From time of first chemotherapy or targeted therapy to time of progression or death（according to RECIST v1.1）
Thoracic Progression Free Survival | up to 5 years
  From time of first chemotherapy or targeted therapy to time of progression or death
Overall Survival | up to 5 years
  From time of first chemotherapy or targeted therapy to date of death

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoxia Zhu, Study Chair — Nanfang Hospital, Southern Medical University
Locations (1):
- Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No